CLINICAL TRIAL: NCT02103023
Title: Intradermal Trivalent Influenza Vaccine in Young Adults, a Double-blind Randomized Controlled Trial
Brief Title: Intradermal Influenza Vaccine in the Young
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Ivan FN Hung, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UW 14-016
Record Dates: First submitted 2014-03-28; First posted 2014-04-03 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Influenza Viral Infections
MeSH Terms: interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ID TIV + imiquimod (Experimental): imiquimod ointment followed by intradermal influenza vaccine
  Interventions: Drug: Imiquimod ointment; Biological: Intradermal influenza vaccine
- ID sham + imiquimod (Sham Comparator): imiquimod ointment followed by sham intradermal influenza vaccine
  Interventions: Drug: Imiquimod ointment
- IM TIV + aq (Active Comparator): aqueous cream followed by intramuscular influenza vaccine
  Interventions: Drug: Aqueous cream; Biological: Intramuscular influenza vaccine
- ID TIV + aq (Active Comparator): aqueous cream followed by intradermal influenza vaccine
  Interventions: Drug: Aqueous cream; Biological: Intradermal influenza vaccine

INTERVENTIONS:
Drug: Imiquimod ointment — 5% 250mg imiquimod ointment
  Other Names: Aldara
  Arms: ID TIV + imiquimod; ID sham + imiquimod
Drug: Aqueous cream — aqueous cream
  Other Names: Aqueous cream BP
  Arms: ID TIV + aq; IM TIV + aq
Biological: Intradermal influenza vaccine — intradermal trivalent influenza vaccine (Intanza15)
  Arms: ID TIV + aq; ID TIV + imiquimod
Biological: Intramuscular influenza vaccine — intramuscular trivalent influenza vaccine (Vaxigrip)
  Arms: IM TIV + aq

SUMMARY:
Influenza poses a heavy burden to our health service. The WHO estimates that seasonal influenza causes 250,000-500,000 deaths worldwide each year. Various strategies including intradermal vaccination and new vaccine adjuvants have been shown to improve immunogenicity. Recently, imiquimod, a synthetic Toll-like receptor 7 (TLR7) agonist useful for the treatment of DNA virus infection, have been shown to improve vaccine immunogenicity against influenza virus in mouse model. The objective of this prospective double-blind randomized controlled trial is to evaluate the effect and safety of topical treatment with imiquimod immediately before intradermal influenza vaccination in healthy young adults.

DETAILED DESCRIPTION:
Influenza poses a heavy burden to our health service. Seasonal, zoonotic and pandemic influenza are constant global threats. The WHO estimates that seasonal influenza causes 250,000-500,000 deaths worldwide each year, with an even higher mortality during the pandemic periods. Moreover zoonotic influenza such as the avian-origin H5N1 and more recently the H7N9 influenza are associated with a much higher mortality than seasonal influenza. Vaccine immunogenicity among elderly individuals is also suboptimal due to immunosenescence. Various strategies including intradermal vaccination and new vaccine adjuvants have been shown to improve immunogenicity.

Recently, imiquimod, a synthetic Toll-like receptor 7 (TLR7) agonist useful for the treatment of DNA virus infection, have been shown to improve vaccine immunogenicity against influenza virus in both mouse model. The objective of this prospective double-blind randomized controlled trial is to evaluate the effect and safety of topical treatment with imiquimod immediately before intradermal influenza vaccination. Our a priori hypothesis is that imiquimod pretreatment would expedite and augment the immunogenicity of influenza vaccination.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients at the age of 18-30 years and given written informed consent
* Subjects must be available to complete the study and comply with study procedures.
* Willingness to allow for serum samples to be stored beyond the study period, for potential additional future testing to better characterize immune response.

Exclusion Criteria:

* Clinically significant immune-related diseases or significant recent co-morbidities
* Inability to comprehend and to follow all required study procedures
* History or any illness that might interfere with the results of the study or pose additional risk to the subjects due to participation in the study
* Have received trivalent influenza vaccine within the same year
* Have a recent history (documented, confirmed or suspected) of a flu-like disease within a week of vaccination.
* Have a known allergy to eggs or other components of the Study Vaccines (including gelatin, formaldehyde, octoxinol, thimerosal, and chicken protein), or history of any anaphylaxis, serious vaccine reactions, to any excipients.
* Have a positive urine or serum pregnancy test within 24 hours prior to vaccination, or women who are breastfeeding.
* Female of childbearing potential, not using any acceptable contraceptive methods for at least 2 months prior to study entry or that do not plan to use acceptable birth control measures during the first 3 weeks after vaccination.
* Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months.
* Have an active neoplastic disease or a history of any hematologic malignancy.
* Have long-term use of glucocorticoids including oral, parenteral or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months. (Nasal and topical steroids are allowed).
* Have a history of receiving immunoglobulin or other blood product within the 3 months prior to vaccination in this study.
* Have known active human immunodeficiency virus (HIV), Hepatitis C infection or autoimmune hepatitis and cirrhosis.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during this study. Unwilling to refuse participation in another clinical study through the end of this study.
* History of progressive or severe neurological disorders Have received any licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to vaccination in this study or plan receipt of such vaccines within 21 days following the second vaccination (only exception being unadjuvanted seasonal influenza vaccines which are allowed until 1 week prior to and after 1 week study vaccinations).
* Axillary temperature ≥ 38°C or oral temperature ≥ 38.5°C within 3 days of intended study vaccination
* Surgery planned during the study period that in the Investigator's opinion would interfere with the study visits schedule
* Have a history of alcohol or drug abuse in the last 5 years.
* Have a history of Guillain-Barré Syndrome. Have any condition that the investigator believes may interfere with successful completion of the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate | Day 7
  Hemagglutination inhibition assay

SECONDARY OUTCOMES:
Seroprotection rate | Day 7
  Hemagglutination inhibition assay
GMT fold increase | Day 7
  Hemagglutination inhibition assay
GMT | Day 7
  Microneutralization antibody assay
Seroconversion rate | Day 21
  Hemagglutination inhibition assay
Seroprotection rate | Day 21
  Hemagglutination inhibition assay
GMT fold increase | Day 21
  Hemagglutination inhibition assay
GMT | Day 21
  Microneutralization antibody assay
Adverse events | Day 7
  Solicited local and systemic adverse reactions monitored from time of vaccination till day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Kwok-Yung Yuen, MD FRCP, Study Chair — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Hung IF, Zhang AJ, To KK, Chan JF, Li P, Wong TL, Zhang R, Chan TC, Chan BC, Wai HH, Chan LW, Fong HP, Hui RK, Kong KL, Leung AC, Ngan AH, Tsang LW, Yeung AP, Yiu GC, Yung W, Lau JY, Chen H, Chan KH, Yuen KY. Topical imiquimod before intradermal trivalent influenza vaccine for protection against heterologous non-vaccine and antigenically drifted viruses: a single-centre, double-blind, randomised, controlled phase 2b/3 trial. Lancet Infect Dis. 2016 Feb;16(2):209-18. doi: 10.1016/S1473-3099(15)00354-0. Epub 2015 Nov 9. PMID 26559482